CLINICAL TRIAL: NCT03948776
Title: Validation of Body Composition Ultrasound for Identification of Sarcopenia and Cachexia in Patients With Heart Failure
Brief Title: Body Composition Ultrasound for Patients With Heart Failure
Status: Completed | Type: Observational
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 13206
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (4):
- Healthy volunteers: Adults without HF or prior heart transplantation
  Interventions: Diagnostic Test: BodyMetrix body composition ultrasound
- Participants in our existing LVAD body composition study: Currently-enrolled LVAD body composition participants, who chose to participate in this study on the same day as a DXA scan already scheduled for study #12026
  Interventions: Diagnostic Test: BodyMetrix body composition ultrasound
- Patients with heart failure, an LVAD or heart transplantation: Any patients with a current diagnosis of HF, with or without an LVAD, or prior HF now status post heart transplantation
  Interventions: Diagnostic Test: BodyMetrix body composition ultrasound
- Inpatients with heart failure, LVAD, heart transplantation: Patients with a current diagnosis of HF, with or without an LVAD, or prior HF now status post heart transplantation, currently admitted as inpatients at Tufts Medical Center. The 6/20/2019 protocol update includes these patients who will participate without a DXA scan (which can only be performed as an outpatient).
  Interventions: Diagnostic Test: BodyMetrix body composition ultrasound only

INTERVENTIONS:
Diagnostic Test: BodyMetrix body composition ultrasound — Investigators will make ultrasound measurements of fat and muscle thickness at 7 positions on the arm, chest wall, and leg (subject's dominant side) using the BodyMetrix BX 2000 ultrasound machine. Clear ultrasound gel will be applied to the skin, a probe placed against the skin, and the fat/muscle thickness measurement made five times at each position. The gel is then wiped away. The images are analyzed by the BodyView Software and estimations of fat and muscle mass calculated. These will be compared to the reference technique of whole-body DXA imaging.
  Groups: Healthy volunteers; Participants in our existing LVAD body composition study; Patients with heart failure, an LVAD or heart transplantation
Diagnostic Test: BodyMetrix body composition ultrasound only — Investigators will make ultrasound measurements of fat and muscle thickness at 7 positions on the arm, chest wall, and leg (subject's dominant side) using the BodyMetrix BX 2000 ultrasound machine. Clear ultrasound gel will be applied to the skin, a probe placed against the skin, and the fat/muscle thickness measurement made five times at each position. The gel is then wiped away. The images are analyzed by the BodyView Software and estimations of fat and muscle mass calculated. For inpatients currently admitted to the hospital, whole-body DXA imaging cannot be performed, as so the only assessment of body composition will be with the ultrasound.
  Groups: Inpatients with heart failure, LVAD, heart transplantation

SUMMARY:
This study aims to determine whether skeletal muscle ultrasound is a useful technique for measuring low muscle mass in patients with heart failure (HF). Muscle wasting and abnormal muscle quality has been identified in patients with advanced HF and may contribute to patients' physical limitations. However assessments of body composition for patients with HF currently rely on the research tool of dual X-ray absorptiometry (DXA) for measurements of skeletal muscle mass, which is limited by cost, use of radiation, and the need for patients to be transported to the DXA scanner for imaging. Therefore this observational study is designed to validate a new approach that allows a safe and portable assessment of body composition.

DETAILED DESCRIPTION:
The investigators will be recruiting both healthy subjects without HF, as well as subjects with either HF, a left ventricular assist device (LVAD) or cardiac transplantation. This is an observational study to validate the use of the BodyMetrix BX 2000 Pro ultrasound machine for the assessment of body composition, particularly muscle wasting. The ultrasound device received 501(k) designation from the FDA in 2009 for measurement of localized fat and muscle thickness. Participation will last for only one day, with approximately 2 hours of study activity in total:

1. For woman with child-bearing potential, potential participants will be required to undergo a urine pregnancy test prior to DXA imaging.
2. The investigators will record participant age, sex, height, weight and heart failure status.
3. Muscle ultrasound: investigators will make measurements at 7 positions on the arm, chest wall, and leg (participant's dominant side). Clear ultrasound gel will be applied to the skin, a BodyMetrix ultrasound probe placed against the skin, and the muscle thickness measurement made five times at each position. The gel is then wiped away.
4. Whole body dual X-ray absorptiometry (DXA) scan: the DXA scan involves lying on a flat and open scanner for approximately 5 minutes while an X-ray arm passes over the body to form a picture for whole body composition.
5. Handgrip strength: this involves the participant squeezing a handheld machine on three occasions in the dominant hand to measure grip strength.
6. 5 sit-to-stand test: investigators will time how long it takes for the participant to stand up from a seated position five times to assess lower body strength.

ELIGIBILITY:
Inclusion Criteria:

1. Cohort 1: Healthy volunteers:

   * 18+ years
   * No history of heart failure
   * Not pregnant
   * Willing to take a urinary pregnancy test if there is a possibility of pregnancy
   * Able to freely provide informed consent
2. Cohort 2: Participants in our existing left ventricular assist device (LVAD) body composition study (#12026) who consent to undergo skeletal muscle ultrasound the same day as an LVAD body composition study visit that already includes the DXA and handgrip strength procedures:

   • Meet the eligibility criteria outlined in study #12026
3. Cohort 3: Patients with heart failure, an LVAD or heart transplantation

   * 18+ years
   * Not pregnant
   * Willing to take a urinary pregnancy test if there is a possibility of pregnancy

Exclusion Criteria:

1. Patients requiring temporary mechanical circulatory support
2. Pregnant women, or women who report there is a possibility they could be pregnant and decline to complete a pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three study populations will be recruited for this observational validation study:
  Cohort 1: Healthy volunteers Cohort 2: Participants in our existing left ventricular assist device (LVAD) body composition study (#12026) who consent to undergo skeletal muscle ultrasound the same day as an LVAD body composition study visit that already includes the DXA and handgrip strength procedures Cohort 3: Patients with heart failure, an LVAD or heart transplantation Cohort 4: Inpatients with heart failure, an LVAD or heart transplantation, currently admitted to Tufts Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Primary DXA endpoint: fat free mass (FFM) measured by DXA | On study day 1
  This is the fat free mass calculated by whole-body DXA, which is the gold standard for measuring skeletal muscle mass
Primary ultrasound endpoint: FFM measured by BodyMetrix ultrasound | On study day 1
  This is the muscle mass estimation from the BodyMetrix ultrasound device which the investigators are seeking to validate as a method of body composition assessment

SECONDARY OUTCOMES:
Handgrip strength | On study day 1
  Average of 3 handgrip strength measurements in the dominant upper extremity
Sit-to-stand test | On study day 1
  Time (in seconds) for the participant complete 5 sit-to-stands, starting in a seated position on a chair

CONTACTS AND LOCATIONS:
Overall Officials: Amanda R Vest, MBBS, MPH, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perkisas S, Baudry S, Bauer J, Beckwee D, De Cock AM, Hobbelen H, Jager-Wittenaar H, Kasiukiewicz A, Landi F, Marco E, Merello A, Piotrowicz K, Sanchez E, Sanchez-Rodriguez D, Scafoglieri A, Cruz-Jentoft A, Vandewoude M. Application of ultrasound for muscle assessment in sarcopenia: towards standardized measurements. Eur Geriatr Med. 2018 Dec;9(6):739-757. doi: 10.1007/s41999-018-0104-9. Epub 2018 Sep 17. PMID 34674473
- [Background] Abe T, Fujita E, Thiebaud RS, Loenneke JP, Akamine T. Ultrasound-Derived Forearm Muscle Thickness Is a Powerful Predictor for Estimating DXA-Derived Appendicular Lean Mass in Japanese Older Adults. Ultrasound Med Biol. 2016 Sep;42(9):2341-4. doi: 10.1016/j.ultrasmedbio.2016.05.008. Epub 2016 Jun 17. PMID 27321173
- [Background] Abe T, Loenneke JP, Young KC, Thiebaud RS, Nahar VK, Hollaway KM, Stover CD, Ford MA, Bass MA, Loftin M. Validity of ultrasound prediction equations for total and regional muscularity in middle-aged and older men and women. Ultrasound Med Biol. 2015 Feb;41(2):557-64. doi: 10.1016/j.ultrasmedbio.2014.09.007. Epub 2014 Nov 25. PMID 25444689
- [Background] Takai Y, Ohta M, Akagi R, Kato E, Wakahara T, Kawakami Y, Fukunaga T, Kanehisa H. Applicability of ultrasound muscle thickness measurements for predicting fat-free mass in elderly population. J Nutr Health Aging. 2014;18(6):579-85. doi: 10.1007/s12603-013-0419-7. PMID 24950147

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/76/NCT03948776/Prot_SAP_002.pdf